CLINICAL TRIAL: NCT07232238
Title: TRPM2 Gene Polymorphism in Relation to NLRP3 Inflammasome Expression in Vitiligo Patients
Brief Title: TRPM2 Gene Polymorphism, NLRP3 Inflammasome Expression in Vitiligo Patients
Status: Active, not recruiting | Type: Observational
Sponsor: Aswan University (Other)
Responsible Party: Principal Investigator, Mostafa Ahmed Maher Sayed, Principal Investigator / MD Candidate, Aswan University
Other Study IDs: 897/1/24
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-08

CONDITIONS: Vitiligo
Keywords: TRPM2, NLRP3, oxidative stress, inflammasome, genetic polymorphism
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — Peripheral blood samples collected from vitiligo patients and healthy controls for DNA extraction and molecular analysis. Remaining material will be discarded after completion of testing.

GROUPS / COHORTS (2):
- Vitiligo Patients: Participants clinically diagnosed with vitiligo, recruited from the Dermatology Outpatient Clinic, Aswan University Hospital. Peripheral blood samples will be collected for TRPM2 gene and NLRP3 inflammasome analysis.
- Healthy Controls: Age- and sex-matched healthy individuals without autoimmune or inflammatory disorders, recruited as controls. Blood samples will be analyzed similarly for comparison.

SUMMARY:
This study investigates the relationship between Transient Receptor Potential Melastatin 2 (TRPM2) gene polymorphism and Nucleotide-binding oligomerization domain-like receptor protein 3 (NLRP3) inflammasome expression in patients with vitiligo. Vitiligo is a common autoimmune depigmenting disorder characterized by melanocyte destruction associated with oxidative stress and immune dysregulation.

TRPM2 is a calcium-permeable cation channel activated by oxidative stress, while NLRP3 inflammasome activation promotes inflammation through interleukin-1β (IL-1β) and interleukin-18 (IL-18) release. This study aims to evaluate TRPM2 genetic variants, NLRP3 expression levels, and their possible correlation with disease severity measured using the Vitiligo Area Scoring Index (VASI).

DETAILED DESCRIPTION:
Vitiligo is a chronic autoimmune depigmenting disorder characterized by selective loss of melanocytes. Oxidative stress plays a central role in triggering melanocyte damage. Transient Receptor Potential Melastatin 2 (TRPM2) is a calcium-permeable cation channel activated by reactive oxygen species (ROS). Activation of TRPM2 leads to increased intracellular calcium (Ca2+) influx and mitochondrial dysfunction, contributing to melanocyte apoptosis.

The Nucleotide-binding oligomerization domain-like receptor protein 3 (NLRP3) inflammasome is an intracellular multiprotein complex activated by cellular stress signals, including Ca2+ influx, ROS, and mitochondrial injury. NLRP3 activation results in caspase-1 activation and the release of pro-inflammatory cytokines interleukin-1β (IL-1β) and interleukin-18 (IL-18), which further contribute to melanocyte destruction.

Evidence suggests an interaction between TRPM2 activation and NLRP3 inflammasome signaling, particularly under oxidative stress conditions. However, this relationship has not been studied in vitiligo patients. This study investigates TRPM2 gene polymorphism, evaluates NLRP3 expression levels, and explores their association with disease presence and severity.

ELIGIBILITY:
Inclusion Criteria:

- Adult patients (aged 18 years and older) clinically diagnosed with vitiligo, either newly diagnosed or not on treatment for at least 3 months before the study.

Exclusion Criteria:

* Any participant with associated inflammatory disease (such as infections or autoimmune disorders).
* Patients with chronic diseases including cardiac, hepatic, hematologic, or renal disorders, or malignancies.
* Patients who had recent major surgical procedures.
* Patients with segmental vitiligo.
* Vitiligo patients who have received treatment within 3 months prior to the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients with clinically diagnosed vitiligo attending the Dermatology Department at Aswan University Hospital, Egypt, and healthy control participants matched for age and sex.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-10-20 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
TRPM2 gene polymorphism in vitiligo patients | At time of enrollment (single visit)
  Assessment of TRPM2 gene polymorphism by SNP genotyping in blood samples from vitiligo patients and healthy controls. The frequency and distribution of TRPM2 variants will be compared between groups.

SECONDARY OUTCOMES:
NLRP3 inflammasome expression in vitiligo patients | At time of enrollment (single visit)
  Quantification of NLRP3 inflammasome gene expression by real-time PCR (RT-qPCR) in peripheral blood of vitiligo patients and healthy controls. Expression levels will be compared between groups.
Correlation between TRPM2 polymorphism and NLRP3 inflammasome expression | At time of enrollment (single visit)
  Correlation analysis between TRPM2 gene polymorphism and NLRP3 inflammasome expression among vitiligo patients to assess possible functional association.
Association between TRPM2 gene polymorphism and disease severity | At time of enrollment (single visit)
  Comparison of TRPM2 gene polymorphism variants with vitiligo severity measured by Vitiligo Area Severity Index (VASI).
  The Vitiligo Area Scoring Index (VASI) is a validated tool used to quantify vitiligo severity. Scores range from 0 to 100, where higher scores indicate greater disease severity. Assessment is performed at a single study visit.

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa Ahmed Maher, M.B.B.Ch., Principal Investigator — Faculty of Medicine, Aswan University
Locations (1):
- Aswan University Hospital, Aswān, Aswan Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared. Summary results will be available in the final thesis and related publications.

REFERENCES:
- See also: Faculty of Medicine, Aswan University official website. — https://www.aswu.edu.eg/faculty-of-medicine